CLINICAL TRIAL: NCT01464450
Title: PK Study of Oral Rivaroxaban in Healthy Subjects
Brief Title: Pharmacokinetics Study of Oral Rivaroxaban in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100688; RIVAROXNAP1001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Pharmacokinetics; Bioavailability; Healthy Participants
Keywords: Pharmacokinetics; Bioavailability; Healthy Participants
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1: Treatment A - B - C (Active Comparator): Participants will receive a single 20 mg-dose of rivaroxaban as a whole tablet swallowed intact with 70 mL of applesauce and 130 mL of water followed by a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 1 (Treatment A,) followed by a single 20 mg-dose of rivaroxaban crushed and mixed in 70 ml of applesauce, followed by 2 mortar rinses of 65 mL each of water (to ensure delivery of the entire dose) and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 2 (Treatment B) and followed by 20 mL of water via NG tube (to prime and pre-wet the lumen), followed by a single 20 mg-dose of rivaroxaban crushed and suspended in 50 mL of water given via NG tube, followed by 2 mortar rinses of 65 mL each of water and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 3 (Treatment C.)
  Interventions: Drug: Rivaroxaban
- Sequence 2: Treatment A - C - B (Active Comparator): Participants will receive a single 20 mg-dose of rivaroxaban as a whole tablet swallowed intact with 70 mL of applesauce and 130 mL of water followed by a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 1 (Treatment A,) followed by 20 mL of water via NG tube (to prime and pre-wet the lumen), followed by a single 20 mg-dose of rivaroxaban crushed and suspended in 50 mL of water given via NG tube, followed by 2 mortar rinses of 65 mL each of water and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 2 (Treatment C) and followed by a single 20 mg-dose of rivaroxaban crushed and mixed in 70 ml of applesauce, followed by 2 mortar rinses of 65 mL each of water (to ensure delivery of the entire dose) and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 3 (Treatment B.)
  Interventions: Drug: Rivaroxaban
- Sequence 3: Treatment B - C - A (Active Comparator): Participants will receive a single 20 mg-dose of rivaroxaban crushed and mixed in 70 ml of applesauce, followed by 2 mortar rinses of 65 mL each of water (to ensure delivery of the entire dose) and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 1 (Treatment B,) followed by a single 20 mg-dose of rivaroxaban crushed and suspended in 50 mL of water given via NG tube, followed by 2 mortar rinses of 65 mL each of water and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 2 (Treatment C) and followed by a single 20 mg-dose of rivaroxaban as a whole tablet swallowed intact with 70 mL of applesauce and 130 mL of water followed by a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 3 (Treatment A.)
  Interventions: Drug: Rivaroxaban
- Sequence 4: Treatment B - A - C (Active Comparator): Participants will receive a single 20 mg-dose of rivaroxaban crushed and mixed in 70 ml of applesauce, followed by 2 mortar rinses of 65 mL each of water (to ensure delivery of the entire dose) and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 1 (Treatment B,) followed by a single 20 mg-dose of rivaroxaban as a whole tablet swallowed intact with 70 mL of applesauce and 130 mL of water followed by a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 2 (Treatment A) and followed by 20 mL of water via NG tube (to prime and pre-wet the lumen), followed by a single 20 mg-dose of rivaroxaban crushed and suspended in 50 mL of water given via NG tube, followed by 2 mortar rinses of 65 mL each of water and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 3 (Treatment C.)
  Interventions: Drug: Rivaroxaban
- Sequence 5: Treatment C - A - B (Active Comparator): Participants will receive a single 20 mg-dose of rivaroxaban crushed and suspended in 50 mL of water given via NG tube, followed by 2 mortar rinses of 65 mL each of water and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 1 (Treatment C,) followed by a single 20 mg-dose of rivaroxaban as a whole tablet swallowed intact with 70 mL of applesauce and 130 mL of water followed by a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 2 (Treatment A) and followed by and followed by a single 20 mg-dose of rivaroxaban crushed and mixed in 70 ml of applesauce, followed by 2 mortar rinses of 65 mL each of water (to ensure delivery of the entire dose) and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 3 (Treatment B.)
  Interventions: Drug: Rivaroxaban
- Sequence 6: Treatment C - B - A (Active Comparator): Participants will receive a single 20 mg-dose of rivaroxaban crushed and suspended in 50 mL of water given via NG tube, followed by 2 mortar rinses of 65 mL each of water and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 1 (Treatment C,) followed by and followed by a single 20 mg-dose of rivaroxaban crushed and mixed in 70 ml of applesauce, followed by 2 mortar rinses of 65 mL each of water (to ensure delivery of the entire dose) and a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 2 (Treatment B) and followed by a single 20 mg-dose of rivaroxaban as a whole tablet swallowed intact with 70 mL of applesauce and 130 mL of water followed by a liquid meal (100 mL of Osmolite® 1.5 Cal at 0, 0.5, 1, 1.5 and 2 hours after receiving the study drug) in Period 3 (Treatment A.)
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Single 20 mg-dose

SUMMARY:
The primary objective of this study is to learn about the relative bioavailability (the extent to which the drug becomes available to the body) and pharmacokinetics (blood levels) of rivaroxaban in healthy participants after receiving a 20 mg rivaroxaban tablet orally as a whole tablet, crushed and mixed in applesauce, and as a suspension through a Naso-gastric (NG) tube. The relative bioavailability of rivaroxaban may be different when given as a crushed tablet compared with an intact (whole) tablet and when given via an NG tube. The safety and tolerability of rivaroxaban will also be assessed.

DETAILED DESCRIPTION:
This is a single-center, open-label (all people know the identity of the drug), randomized (the study drug is assigned by chance), 3-period, 3-treatment cross over study of the relative bioavailability (the extent to which the drug becomes available to the body) of single dose rivaroxaban given to healthy participants in 3 ways. All participants will be randomly assigned to follow 1 of 6 possible ordered sequences whereby they ultimately receive rivaroxaban as: a whole tablet orally (Treatment A), a crushed tablet mixed in applesauce orally (Treatment B), and a crushed tablet in a water suspension administered via NG tube (Treatment C). Each rivaroxaban treatment will be taken with food (a standardized liquid meal).

Participants will be randomly assigned into one of the following 6 sequences:

* Sequence 1: Treatment A - Treatment B - Treatment C
* Sequence 2: Treatment A - Treatment C - Treatment B
* Sequence 3: Treatment B - Treatment C - Treatment A
* Sequence 4: Treatment B - Treatment A - Treatment C
* Sequence 5: Treatment C - Treatment A - Treatment B
* Sequence 6: Treatment C - Treatment B - Treatment A.

It is expected that a total of 9 participants will be randomly assigned into each sequence. Each single-dose treatment period will be followed by a washout period (period when receiving no treatment) of sufficient length to ensure absence of drug carry over from one treatment period to the next.

The study will enroll approximately 54 participants to achieve 42 completed participants.

The study will consist of a screening phase (no longer than 21 days before entering the clinical research facility on the day before starting the study drug), randomly assigned to 1 of 6 sequences, and an open-label treatment phase consisting of 3 treatment periods (4 days for each treatment) separated by a washout period of 6-14 days between rivaroxaban administrations in each treatment periods.

Participants will be admitted to the study unit in the morning of the day before the giving of the first dose of study drug (Day -1). Study drug will be given in the morning of the first day of each treatment period (Day 1), followed by a standard Osmolite® 1.5 Cal (Abbott Laboratories) liquid meal.

Participants will receive study drug in the morning and Osmolite® 1.5 Cal will be given as the breakfast meal. Osmolite® 1.5 Cal is a standardized source of balanced nutrition for patients requiring low-residue meals via a feeding tube or orally and/or who may have limited volume tolerance or fluid restrictions. An Osmolite® 1.5 Cal meal includes 1.5 calories/mL overall, and 62.7 g of protein/L. Participants can have a regular meal 3 or more hours after the Osmolite® 1.5 Cal meal.

Each treatment period will be followed by a 6 to 14 day washout period. The washout period will start after the giving of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, clinical laboratory tests, vital signs, and 12-lead Electrocardiogram (ECG) performed at screening; Non-smoker for at least 3 months before screening; Women must be postmenopausal, surgically sterile or practicing a highly effective method of birth control; Men must agree to use birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug; Body Mass Index (BMI) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg.; Be willing and able to adhere to the prohibitions and restrictions specified in this protocol;

Exclusion Criteria:

* History of or current clinically significant medical illness; Allergies, hypersensitivity, or intolerance to any component of rivaroxaban or its excipients or to Osmolite® 1.5 Cal; Contraindications to the use of anticoagulant (a drug used to thin blood) therapy (eg, bleeding diathesis, history of gastrointestinal (GI) bleeding within 1 year or coagulopathy); History of any disorder known to increase the risk of bleeding; Hepatic dysfunction and/or elevated serum transaminases; Clinically relevant hepatosplenomegaly as determined by the study investigator; Renal insufficiency; History of malignancy within 2 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence); Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 1 month before the planned first dose of study drug; Any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments; Had major surgery, (eg, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or planned surgery during the time the subject is expected to participate in the study or within 12 weeks after the last dose of study agent is given; Uses any prescription or nonprescription medication (including vitamins and herbal supplements), except for (with restrictions) acetaminophen, oral contraceptives, and hormonal replacement therapy (stable dose) within 14 days before the first dose of the study drug is scheduled up to be given up to the End of Study/Early Withdrawal; History of drug or alcohol abuse within the past 2 years or a positive test for drugs of abuse at screening; Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before receiving the study drug or intention or donation of blood or blood products within 1 month before receiving the study drug, during the study or within 1 month after the completion of the study; Unable to swallow solid, oral dosage forms whole with the aid of water, crushed forms mixed with apple sauce or tolerate placement of a NG tube for delivery of drug suspension; Has a history of testing positive for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rivaroxaban plasma concentrations | Approximately 30 days

SECONDARY OUTCOMES:
The number of patients with adverse events reported | Up to approximately 60 days
Change from baseline in coagulation tests (prothrombin time [PT] and partial thromboplastin time [PTT]) | Baseline and at approximately 47 days
Change from baseline in Electrocardiograms (ECGs) | Baseline and at approximately 47 days
Number of participants with abnormal vital signs | Baseline and at approximately 10 days, 20 days and 30 days
Number of participants with changes in physical examinations | Baseline and at approximately 10 days, 20 days and 30 days
Urine Drug Screen | Baseline and at approximately 10 days and 20 days
Change from baseline in clinical lab assessments (chemistry, hemotology) | Baseline and at approximately 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Neptune City, New Jersey, United States